CLINICAL TRIAL: NCT02258620
Title: Prevention and Comparison of Different Forms of Administration of Nitrates in the Risk of Radial Spasm During Coronary Angiography.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, José Castro, Chef de Clinique, Brugmann University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUB-SAR
Record Dates: First submitted 2014-09-26; First posted 2014-10-07 (Estimated); Last update posted 2014-10-07 (Estimated); Status verified 2014-10

CONDITIONS: Coronaropathy
MeSH Terms: interventions — Isosorbide; Nitroglycerin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- dinitrate isosorbide (intra venous) (Experimental): dinitrate isosorbide by continuous intra venous injection (1 à 5 mg/h)
  Interventions: Drug: dinitrate isosorbide
- dinitrate isosorbide (intra arterial) (Experimental): dinitrate isosorbide 5 mg by direct administration intra arterial
  Interventions: Drug: dinitrate isosorbide
- nitroglycerine (transdermic) (Experimental): nitroglycerine dermal patch15 mg/24h soit 67,2 mg/21 cm2
  Interventions: Drug: nitroglycerine

INTERVENTIONS:
Drug: dinitrate isosorbide — dinitrate isosorbide (cedocard*) by continuous intra venous (1 to 5 mg/h) dinitrate isosorbide (cedocard*) 5 mg by intra arterial direct in the sheat
  Arms: dinitrate isosorbide (intra arterial); dinitrate isosorbide (intra venous)
Drug: nitroglycerine — nitroglycerine dermal patch 15 mg/24h : 67,2 mg/21 cm2
  Arms: nitroglycerine (transdermic)

SUMMARY:
The radial approach for a coronary angiography is currently adopted by several centers because of its simplicity. The radial artery spasm is the main inconvenient. Nitrates in intra-arterial have been widely studied in prevention of this spasm. No studies have compared the different routes of administration of nitrates as a patch and a continuous intravenous injection.

DETAILED DESCRIPTION:
The radial approach is favored for coronary angiography due of several advantages: reduction of local bleeding risk, even in the most hemorragiparic situations, decreased downtime and time reduction of hospitalization, improved patient ulterior comfort. However, this approach is subject to an immediate major complication that is the radial artery spasm (RAS) which, according to the criteria used, has an average incidence of 30%. The administration of a vasodilator just before coronary angiography procedure enables an increase of the radial artery diameter and thus a decrease of friction probes. Theoretically this prevents the occurrence of the RAS.

The literature re-counts several vasodilator product tests (DN calcic blocker, magnesium sulfate, alpha-adrenergic antagonist ...) and various routes of administration (direct intravenous route (IV), subcutaneous injected route, direct intra-arterial route (IA)). Overall intra-arterial DN appears to be more efficient. The downside is a brief, painful thermal sensation but intense and notably unpleasant. IV injection is better tolerated but it was a direct injection and without proof of its superiority over IA. The para-radial subcutaneous injection has only been studied to facilitate access to the radial artery. The investigators randomized study compares, for the first time, the effectiveness of the transdermal administration of trinitrine (D) and continuous intravenous of dinitrate isosorbide (V) to dinitrate isosorbide intraarterial (A) standard.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 ans.
* Patients with hemodynamic stability.
* Patients informed consent was signed by each individual. The study obtained approval from the local ethics committee.

Exclusion Criteria:

* 'Test d'Allen' negative
* Pregnancy.
* STEMI
* Hemodynamic Instability : PAS < 100 mmHg, FC > 100 bpm, tachycardia uncontrollable.
* Allergy of nitrates.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2013-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Radial artery diameter | Day of administration
  With the help of an arterial doppler, measure of the radial artery diameter after injection of dinitrate isosorbide at the beginning and at the end of the procedure (objective measure)
Probe friction | Day of administration
  Probe friction, as experienced by the operator (subjective measure)
Pain | Day of administration
  Pain felt by the patient in the forearm (subjective measure)
Radial artery occlusion | 3 months post procedure
  Evaluation of the radial artery occlusion 3 months post procedure

CONTACTS AND LOCATIONS:
Overall Officials: José Castro, MD, Principal Investigator — CHU-Brugmann
Locations (1):
- CHU-Brugmann, Brussels, Belgium